CLINICAL TRIAL: NCT03932032
Title: Targeting Attention Orienting to Social Threat to Reduce Social Anxiety in Youth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH119299 (NIH)
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Social Anxiety Disorder of Childhood

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Bias Modification Treatment (Experimental): Attention Bias Modification Treatment is a computer-based attention training program.
  Interventions: Behavioral: Attention Bias Modification Treatment
- Neutral Control Task (Sham Comparator): Neutral Control Task uses the same computer-based format as Attention Bias Modification Treatment, but includes only neutral stimuli and does not train attention.
  Interventions: Behavioral: Neutral Control Task

INTERVENTIONS:
Behavioral: Attention Bias Modification Treatment — At each of eight sessions, participants complete 160 computer administered trials wherein a pair of threatening stimuli and neutral stimuli is presented simultaneously and then followed immediately by a probe. The probe always replaces the neutral stimulus and never replaces the threatening stimulus. The intervention is based on the idea that attention can be shaped via repetitive computer based training methods, and training attention toward neutral stimuli will lead to a reduction in social anxiety.
  Arms: Attention Bias Modification Treatment
Behavioral: Neutral Control Task — At each of eight sessions, participants complete 160 computer administered trials wherein a pair of neutral stimuli is presented simultaneously and then followed immediately by a probe. NCT matches ABMT on duration, format, and number of trials, but does not engage attention to social threat and does not train attention.
  Arms: Neutral Control Task

SUMMARY:
This two-site study is a test of Attention Bias Modification Treatment (ABMT) among 260 youths ages 10 to 14 years with social anxiety disorder. One-half of participants will receive 8 sessions of computer administered ABMT and the other half of participants will receive 8 sessions of computer administered Neutral Control Task (NCT). The investigators hypothesize that a biomarker of attention to social threat measured using electroencephalography (EEG) and ratings of social anxiety severity will be lower in participants who receive ABMT compared to participants who receive NCT.

ELIGIBILITY:
Inclusion Criteria:

* Be between ages 10 and 14 years
* meet DSM5 criteria for a diagnosis of Social Anxiety Disorder
* presence of any coexisting psychiatric diagnoses must be of lesser severity than Social Anxiety Disorder
* have no current psychotropic medication other than a stable dose of stimulant or non-stimulant medication for coexisting ADHD

Exclusion Criteria:

* meet DSM5 criteria for Autism Spectrum Disorder, Intellectual Disability, Bipolar Disorder, Tourette's Disorder, Psychotic Disorders, or Substance Use Disorders
* show high likelihood of hurting self or others
* be a victim of undisclosed abuse requiring investigation/ supervision by the Department of Social Services
* have an uncorrected vision or physical disability that interferes with the ability to click a mouse button rapidly and repeatedly
* have a history of neurological illness, including seizures/epilepsy, or head injury with loss of consciousness > 5 minutes

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
P1 amplitude elicited in the dot-probe task | post-intervention (within one week of completing the final treatment session)
  Posttreatment event related potential amplitude elicited during the emotional faces dot probe task. The investigators will focus specifically on the P1 amplitude time-locked to the onset of facial stimuli in the dot probe task. P1 amplitude will be measured using EEG methodology.
P1 amplitude elicited in the dot-probe task | Follow-up (six months after completing the final treatment session)
  Follow-up P1 event related potential amplitude elicited during the emotional faces dot probe task. The investigators will focus specifically on the P1 amplitude time-locked to the onset of facial stimuli in the dot probe task. P1 amplitude will be measured using EEG methodology.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale for Children and Adolescents | post-intervention (within one week of completing the final treatment session)
  posttreatment clinician rating of youth social anxiety symptom severity over the past 7 days. The name of the measure is the Liebowitz Social Anxiety Scale for Children and Adolescents. It is a clinician rated measure of the severity of youths' social anxiety symptoms. Total scores range from 0 to 144, with higher scores representing more severe social anxiety.
Liebowitz Social Anxiety Scale for Children and Adolescents | Follow-up (six months after completing the final treatment session)
  Follow-up clinician rating of youth social anxiety symptom severity over the past 7 days. The name of the measure is the Liebowitz Social Anxiety Scale for Children and Adolescents. It is a clinician rated measure of the severity of youths' social anxiety symptoms. Total scores range from 0 to 144, with higher scores representing more severe social anxiety.
Screen for Child Anxiety Related Emotional Disorders - Parent Version at posttreatment | 7 days
  posttreatment parent rating of youth social anxiety symptom severity over the past 7 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P). The SCARED-P is a parent rated measure of the severity of youths' anxiety symptoms, including social anxiety. Total scores on the SCARED-P range from 0 to 82, with higher scores representing more severe anxiety.
Screen for Child Anxiety Related Emotional Disorders - Parent Version at Follow up | 7 days
  follow up parent rating of youth social anxiety symptom severity over the past 7 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P). The SCARED-P is a parent rated measure of the severity of youths' anxiety symptoms, including social anxiety. Total scores on the SCARED-P range from 0 to 82, with higher scores representing more severe anxiety.
Screen for Child Anxiety Related Emotional Disorders - Child Version at posttreatment | 7 days
  posttreatment child rating of youth social anxiety symptom severity over the past 7 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C). The SCARED-C is a child rated measure of the severity of youths' anxiety symptoms, including social anxiety. Total scores on the SCARED-C range from 0 to 82, with higher scores representing more severe anxiety.
Screen for Child Anxiety Related Emotional Disorders - Child Version at Follow-Up | 7 days
  Follow up child rating of youth social anxiety symptom severity over the past 7 days. The name of the measure is the Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C). The SCARED-C is a child rated measure of the severity of youths' anxiety symptoms, including social anxiety. Total scores on the SCARED-C range from 0 to 82, with higher scores representing more severe anxiety.

OTHER OUTCOMES:
State Anxiety before and after a Speech Task | post-intervention (within one week of completing the final treatment session)
  posttreatment State-Trait Anxiety Inventory for Children - State Subscale (STAIC-S) administered before and after a 3-minute speech task.
State Anxiety before and after a Speech Task | Follow-up (six months after completing the final treatment session)
  Follow-up State-Trait Anxiety Inventory for Children - State Subscale (STAIC-S) administered before and after a 3-minute speech task.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy W Pettit, PhD, Principal Investigator — Florida International University; Wendy K Silverman, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Child Study Center Program for Anxiety and Mood Disorders, New Haven, Connecticut
  - Florida International University Center for Children and Families, Miami, Florida